CLINICAL TRIAL: NCT06770751
Title: Family Involvement in the Intensive Care Unit: a Prospective Cohort Study Exploring Its Effects on Sedation Dosages, Delirium, Ventilator-Free Days, and Length of Stay.
Brief Title: Family Involvement in ICU
Status: Recruiting | Type: Observational
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Oguzhan Kayhan, Medical Doctor, Lecturer, Istanbul University - Cerrahpasa
Other Study IDs: 2024/231
Record Dates: First submitted 2025-01-08; First posted 2025-01-13 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2025-01

CONDITIONS: Intensive Care Patients; Relatives; Delirium in the Intensive Care Unit; Sedatives; Family
Keywords: Intensive care patients; relatives; Delirium in the intensive care unit; Sedatives

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Short involvement of family: A group where relatives spend up to 2 hours with patients and are involved in their care.
- Long involvement of family: A group where relatives spend more than 2 hours with patients and are involved in their care.

SUMMARY:
The aim of this prospective cohort study was to investigate the effect of the time spent with relatives of patients treated in a tertiary intensive care unit on patient outcomes.

The main question it aimed to answer was:

Does spending more time with relatives of patients in intensive care result in lower sedative agent requirements? Does spending more time with relatives of patients in intensive care result in less delirium, fewer ventilator days, and shorter ICU stays?

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 and over.
* Patients with at least one family member actively involved in the care process in the ICU.

Exclusion Criteria:

* Patients with pre-existing cognitive impairment or dementia.
* Patients with severe traumatic brain injury.
* Patients with an expected mortality in the ICU of more than 80%.
* Absence of family members for patients admitted to the ICU.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients in a tertiary intensive care unit of a university hospital
Sampling Method: Non-Probability Sample
Enrollment: 122 (Estimated)
Dates: Start 2025-01-13 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-08-15 (Estimated)

PRIMARY OUTCOMES:
Sedative dose | Each patient will be evaluated and recorded daily up to first 4 weeks of their stay in ICU.
  It is the average daily dose of sedative drugs used by a patient. It will be calculated for each sedative drug. It will be calculated by dividing all doses taken by the number of days of hospitalization.

SECONDARY OUTCOMES:
Delirium | Each patient will be evaluated and recorded daily up to first 4 weeks of their stay in ICU.
  Each patient will be assessed for delirium every day during their hospitalization. CAM-ICU scoring will be used for assessment. The average number of delirium days for each patient will be found by dividing the number of days they were in delirium by the total number of days they were in hospital.
Ventilatory days | Each patient will be evaluated and recorded daily up to first 4 weeks of their stay in ICU.
  For each patient, the number of days they are on a ventilator will be calculated as a percentage of their length of stay. For each patient, the days they receive invasive ventilation will be divided by the number of days they are treated in the intensive care unit to calculate the percentage.
Stay in intensive care unit | Each patient will be evaluated and recorded daily up to first 4 weeks of their stay in ICU.
  The length of time each patient stays in intensive care will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Oktay Demirkiran, Professor, Study Director — İstanbul University - Cerrahpaşa, Cerrahpaşa Medical Faculty; Oguzhan Kayhan, Principal Investigator — İstanbul University - Cerrahpaşa, Cerrahpaşa Medical Faculty
Locations (1):
- Cerrahpaşa Medical Faculty, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Ethics committee approval was not obtained for sharing patient data with an international database.